CLINICAL TRIAL: NCT01259466
Title: Internet-Administered Smoking Cessation Treatment for Overweight and Obese Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Marney A. White, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1001006181
Record Dates: First submitted 2010-11-11; First posted 2010-12-14 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Smoking Cessation; Overweight; Obesity
Keywords: Smoking cessation; Overweight; Obesity; Internet treatment
MeSH Terms: conditions — Smoking Cessation; Overweight; Obesity | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral + Nicotine Patch (Experimental): Cognitive Behavioral Therapy + Nicotine Replacement Patch
  Interventions: Drug: Nicotine patch
- Health Education + Nicotine Patch (Active Comparator): Health Education + Nicotine Replacement Patch
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch — Transdermal Nicotine Replacement Therapy - 21 mg daily for 10 weeks
  Other Names: Nicotine replacement

SUMMARY:
This project will be a randomized clinical trial testing the efficacy of an internet-administered smoking cessation treatment for overweight and obese smokers. Research on internet-administered behavioral treatments for smoking cessation has found that compared to control treatments (e.g., self-help materials), cessation rates in internet-administered treatments are significantly higher. Research testing the applicability of these treatments to overweight and obese individuals has not yet been conducted. Given that a substantial portion of smokers are also overweight and at elevated cardiovascular risk, there is a need for directed treatment efforts for this group. The current trial proposes to be the first to test the effectiveness of internet-administered smoking cessation treatment for overweight and obese (BMI≥25) smokers. Adult participants will be randomized to receive 12 weeks of internet-administered treatment consisting of either: a) standard smoking cessation treatment with general health education, or b) standard smoking cessation treatment with cognitive behavioral therapy (CBT) for weight concerns. Participants in both conditions will receive open-label treatment with the 21 mg transdermal nicotine patch.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 10 or more cigarettes per day
* Regular access to the internet
* BMI>=25

Exclusion Criteria:

* Type I diabetes or Type II diabetes requiring medication
* Alcohol or drug dependence within the past year
* Females with current pregnancy or breastfeeding or intention to become pregnant within the next 12 months
* Uncontrolled hypertension
* Severe chronic obstructive pulmonary disease
* Use of an investigational drug within 30 days or current participation in another clinical trial
* Current use of tobacco products other than cigarettes or use of marijuana
* Use of nicotine replacement therapy, clonidine, varenicline, bupropion, or nortriptyline within the month prior to enrollment
* Use of a medication that might affect weight or appetite
* History of allergic reactions to adhesives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marney A White, PhD, MS, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Treatment + Nicotine Replacement; Health Education + Nicotine Replacement: Nicotine patch: Transdermal Nicotine Replacement Therapy - 21 mg daily for 10 weeks
Period: Overall Study
Arm/Group | Cognitive Behavioral Treatment + Nicotine Replacement | Health Education + Nicotine Replacement
Started | 27 | 27
Completed | 26 | 18
Not Completed | 1 | 9
Not completed — Withdrawal by Subject | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Treatment + Nicotine Replacement | Health Education + Nicotine Replacement | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.6) | 45.4 (9.6) | 45.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Verified Smoking Cessation (Abstinence)
Description: Continuous abstinence during the last 14 days of treatment, confirmed by biologically verified abstinence (CO level <10ppm)
Time Frame: Post-treatment (12-weeks)
Measure: Number; unit: participants
Arm/Group | Cognitive Behavioral Treatment + Nicotine Replacement | Health Education + Nicotine Replacement
Number analyzed (Participants) | 27 | 27
participants | 7 | 5

2. Secondary Outcome: Percent Weight Change
Description: % Weight change: ((post-treatment weight - pre-treatment weight)/ pre-treatment weight) * 100
Time Frame: Post-treatment (12 weeks)
Measure: Mean (Standard Deviation); unit: Percent weight change
Arm/Group | Cognitive Behavioral Treatment + Nicotine Replacement | Health Education + Nicotine Replacement
Number analyzed (Participants) | 26 | 18
Percent weight change | 1.47 (2.9) | 1.79 (2.8)

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Treatment + Nicotine Replacement | Health Education + Nicotine Replacement
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No